CLINICAL TRIAL: NCT06761508
Title: Comparison of Different Visual Aids in Enhancing Community Awareness and Promoting Behavioral Change in the Prevention of Hypertension in Anambra State,Nigeria
Brief Title: Comparing of Different Visual Aids Like Video,info-graphics and Pamphlets in Enhancing Community Awareness and Promoting Behavioral Change Towards the Prevention of Hypertension in Basilica of the Most Holy Trinity Onitsha Anambra State,Nigeria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Ottiwu Perpetua Chidiogor, principal investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MH/COMM/523/VOL.111
Record Dates: First submitted 2024-12-15; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
Keywords: Behavioural change in hypertension prevention
MeSH Terms: conditions — Hypertension | interventions — Clinical Trials as Topic

STUDY DESIGN:
Intervention Model Description: This is 3-arm, prospective, parallel (1:1:1), randomized controlled trial. A convenience sampling of registered persons who visit Basilica of the Most Holy Trinity in Onitsha, Anambra State, southeastern Nigeria for regular mass and forums on Sunday. Based on G Power, the total estimated sample size is 81. With proportionate stratification, the number of members required for each stratum of 90 catholic men, 450 catholic women, and 100 catholic youth is 12, 57, and 12, respectively. The participants will be randomly assigned from each stratum to the 3-arms (video, cartoon, pamphlet) based on balloting (draw lots).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- intervention group using video (Other): Administration of video to the first intervention group
  Interventions: Behavioral: Intervention study for Arm one using video
- intervention group using infographics (Other): Administration of infographics to the second arm of the intervention group
  Interventions: Behavioral: intervention 2:using infographics
- control group using pamphlet (Other): Administration of pamphlet to the control groups
  Interventions: Behavioral: intervention 3: use of pamphlet

INTERVENTIONS:
Behavioral: Intervention study for Arm one using video — A 3 Arm randomized control trial, using video as the first Arm of intervention to assess the behaviour change of the community in hypertension prevention.
  Arms: intervention group using video
Behavioral: intervention 2:using infographics — A 3 Arm randomized control trial,that involves the use of infographics in Arm to assess the behaviour change of the community in hypertension prevention.
  Arms: intervention group using infographics
Behavioral: intervention 3: use of pamphlet — A 3 Arm randomized control trial,that contains the use of pamphlet for the 3rd Arm which is the control group to assess the behaviour change of the community in hypertension prevention.
  Arms: control group using pamphlet

SUMMARY:
The goal of this observational study is to assess different level of enhanced awareness and behavioral change of adults over the age of 35 who will be educated using video,infographic and pamphlet for the interval of one month

ELIGIBILITY:
Inclusion Criteria:

* Adults age over 35 years old
* Who does not know his/her blood pressure status within the last 6 months (The person who does not know he or she has a hypertension or not.)
* Who agree to participate

Exclusion Criteria:

* Who cannot come to the church 4 weeks later after the intervention.
* Known hypertensive patients

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Behavioural change in hypertension prevetion | One month
  Behaviour changes within 1 month related to education
  - Asking what kind of behaviour change occurred during 1 month Percentage caculation of participants who had behaviour change Each arm: Number of person who changed their behaviour/total number of participants in the arm

SECONDARY OUTCOMES:
Change in the awareness level of participants from baseline after 4 week | 4 weeks
  - Awareness check: Using the Health belief model-The researchers-developed questionnaire:How much they are motivated (pre and post comparison)

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate School of Biomedical and Health Sciences Hiroshima University, Kasumi 1-2-3 Minami-ku, Japan, Nigeria

IPD SHARING:
Plan to Share IPD: No
To ensure confidentiality